CLINICAL TRIAL: NCT02869113
Title: Evaluation of the Stinging Potential of Sunscreen Products in Human Eyes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 18067
Record Dates: First submitted 2016-08-03; First posted 2016-08-16 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Sunscreen Agents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sunscreen agent A + control (Experimental): Application of control and test product into one of the subjects two eyes.
  Interventions: Drug: BAY98751 (Y65-110); Drug: Standard shampoo mixture (Control)
- Sunscreen agent B + control (Experimental): Application of control and test product into one of the subjects two eyes.
  Interventions: Drug: BAY 98751 (Y65-102); Drug: Standard shampoo mixture (Control)
- Sunscreen agent C + control (Experimental): Application of control and test product into one of the subjects two eyes.
  Interventions: Drug: BAY 98751 (Y65-106); Drug: Standard shampoo mixture (Control)

INTERVENTIONS:
Drug: BAY98751 (Y65-110) — 10 µL in one eye
  Arms: Sunscreen agent A + control
Drug: BAY 98751 (Y65-102) — 10 µL in one eye
  Arms: Sunscreen agent B + control
Drug: BAY 98751 (Y65-106) — 10 µL in one eye
  Arms: Sunscreen agent C + control
Drug: Standard shampoo mixture (Control) — 10 µL in other eye

SUMMARY:
The objective of this study was to compare the human eye stinging potential of experimental formulas and an industry standard shampoo mixture. The study was conducted under the supervision of a Board Certified Ophthalmologist.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged 18 to 60 years
* No medical conditions of the eyes as determined by the subjects' medical history and confirmed by ophthalmologist
* Subjects do not wear contact lenses or, if he/she does wear contact lenses, is willing to refrain from wearing these during the day of and day after the study
* Subject is willing to have the test materials instilled into the eyes and follow all protocol requirements
* Subject is willing to refrain from using false eyelashes of any type or any topical prescription, OTC or cosmetic products on their eyes, eyelids, eyelashes or the peri-orbital areas of the face on the day of the study.
* Subjects should refrain from use of make-up on testing day

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2015-01-23 (Actual); Primary Completion 2015-01-24 (Actual); Study Completion 2015-01-24 (Actual)

PRIMARY OUTCOMES:
Subjective discomfort in the eye was assessed based on questions by an Ophthalmologist to the subject using a 5-category intensity scale | up to 24 hours
Tearing/Lacrimation was assessed by the Ophthalmologist using a 5-category assessment score | up to 24 hours
Objective inflammation was assessed by the Ophthalmologist using a 5-category assessment score | up to 24 hours
Post installation eye effects were assessed using a 5-category intensity score | up to 24 hours

SECONDARY OUTCOMES:
Number of adverse events as a measure of safety and tolerability | at 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- St. Petersburg, Florida, United States